CLINICAL TRIAL: NCT04940312
Title: A Randomized Study to Investigate the Effects of Individualized App-based Coaching on Physical Activity and Myocardial and Vascular Function of Patients with Heart Failure and Preserved Ejection Fraction Compared to Standard Care
Brief Title: MyoMobile Study: App-based Activity Coaching in Patients with Heart Failure and Preserved Ejection Fraction
Acronym: MyoMobile
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Bayer (Industry); McRoberts B.V. (Unknown); Umana Medical Technologies Ltd. (Unknown); International Business Machines (IBM) (Industry)
Responsible Party: Principal Investigator, Philipp Wild, MD, MSc, Univ.-Prof. Dr. med., University Medical Center Mainz
Other Study IDs: UMCM-2020EPI06
Record Dates: First submitted 2021-02-03; First posted 2021-06-25 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Heart Failure, Diastolic
Keywords: Heart failure with preserved ejection fraction (HFpEF); Activity coaching; Smartphone App; Systems Medicine; Clinical Epidemiology
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
  * Serum
  * Plasma (EDTA, citrated, heparinized)
  * DNA
  * RNA Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Usual Care Group: Individuals with heart failure receiving standard medical care
  Interventions: Behavioral: No Intervention: Observational Cohort
- Intervention Group 1 (pedometer-monitoring only): Individuals with heart failure receiving a pedometer for measurement of daily step count
  Interventions: Behavioral: Intervention Group 1
- Intervention Group 2 (app-based coaching): Individuals with heart failure receiving an individualized, app-based physical activity coaching on the basis of pedometer-based assessment of daily step count
  Interventions: Behavioral: App-based physical activity coaching

INTERVENTIONS:
Behavioral: App-based physical activity coaching — Individualized app-based coaching via a smartphone
  Groups: Intervention Group 2 (app-based coaching)
Behavioral: No Intervention: Observational Cohort — no Intervention
  Groups: Usual Care Group
Behavioral: Intervention Group 1 — pedometer-based tracking of physical activity
  Groups: Intervention Group 1 (pedometer-monitoring only)

SUMMARY:
The MyoMobile study is a single-center, randomized, controlled three-armed cohort study with prospective data collection to investigate the effect of a personalized mobile health intervention compared to usual care on the physical activity levels in patients with heart failure and preserved ejection fraction.

DETAILED DESCRIPTION:
Heart failure (HF) affects more than 15 million people in Europe and represents the leading cause of hospitalization. The prevalence of HF is increasing, which has been attributed to an ageing population with subsequently higher prevalence of predisposing risk factors (e.g. arterial hypertension, type-2-diabetes, obesity), a better survival, and more effective treatment of precursors (e.g. myocardial infarction). In the community, heart failure with preserved ejection fraction (HFpEF) is the most common HF phenotype. Currently, the benefit of medical therapies is limited to patients with heart failure with reduced ejection fraction (HFrEF) only, whereas no specific medical therapy is currently approved for patients with HFpEF.

In HF patients, physical inactivity and a sedentary lifestyle lead to disease progression and increased mortality, and an increase of physical activity is positively correlated with improved outcome. Guidelines from the Heart Failure Society of America recommend at least 30 minutes of moderate-intensity activity for ≥ 5 days/week (i.e. at least 150 min/week). Unfortunately, exercise recommendations are poorly implemented in daily clinical practice and even patients enrolled in supervised exercise training programs have been reported to show low adherence.

The MyoMobile study has been designed to assess the effect of a 12-week, app-based coaching program on physical activity in patients with HFpEF. Physical activity including daily step count will be assessed by accelerometry and, in addition, a pedometer will be used to measure the daily step count and provide direct feedback to the patient. Accelerometers provide an objective and continuous assessment of physical activity during patients' daily life over longer periods and may therefore reflect the true effect of the activity coaching intervention on physical activity more accurately than intermittent supervised exercise tests such as the six minute walk test. These efforts are complemented by a comprehensive (sub)clinical and molecular characterization of HFpEF patients at baseline and after the follow-up period of 12 weeks. In order to evaluate the potential effect of awareness for physical activity and of surveillance, due to participants wearing a pedometer throughout the study period, two intervention groups will be investigated. This will allow for the effect of an individualized, app-based coaching intervention, compared to standard care in patients with HFpEF, to be deciphered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Diagnosis of HFpEF

  * LVEF > 40% by any imaging modality at screening within 4 months prior to study entry
  * Current HF symptoms as defined as presence of dyspnea according to New York Heart Association [NYHA] functional class I to III at screening visit
  * Stable HF treatment for at least 4 weeks prior to screening
  * At least one of the following 3 criteria need to be fulfilled: (1) NT-proBNP ≥ 300pg/ml; (2) Hospitalization for HF within the past 12 months; (3) Symptom(s) of HF requiring treatment with diuretic(s) for at least 30 days prior to screening visit
* Wearing time of the physical activity monitor for at least 4 days during the baseline assessment
* Average daily step count during baseline assessment ≥ 1,000 steps per day and < 10,000 steps per day

Exclusion Criteria:

* Acute decompensated HF requiring augmented therapy with diuretic agents, vasodilator agents, and/or inotropic drugs
* Participants who are non-ambulatory managed or use mobility assistive devices such as motorized devices or wheelchairs
* Acute coronary syndrome (including myocardial infarction), cardiac surgery, other major cardiovascular surgery or urgent percutaneous coronary intervention (PCI) within 3 months prior to visit 1 or an elective PCI within 30 days after study enrolment
* Probable alternative diagnoses that in the opinion of the investigator account for the patient's HF symptoms (i.e., dyspnea, fatigue)
* Participants with physical activity impairment primarily due to conditions other than HF such as:

  * Participants unwilling or unable to wear or to operate study measurement devices for the phases required
  * Exertional angina
  * Inflammatory or degenerative joint disease
  * Peripheral vascular disease
  * Neurologic disease affecting activity or mobility (e.g. peripheral neuropathy)
  * Foot ulcer (e.g. diabetic foot syndrome)
  * Prosthetic limbs
* Current chemotherapy and/or radiation therapy for treatment of active cancer
* Medical or psychological conditions that would jeopardize an adequate and orderly conduct or completion of the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with an age of 45 years or older with a diagnosis of heart failure with preserved ejection fraction (HFpEF)
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Average daily step count (all groups) | 12 weeks
  The primary efficacy endpoint is the change in average daily step count between the baseline phase (mean of data collected during the period prior to randomization) and the end of the intervention (mean of data collected during week 12) comparing standard care to a 12-week individualized app-based activity coaching

SECONDARY OUTCOMES:
Difference in E/E' ratio (change from baseline to 12-week follow-up) | 12 weeks
  Difference in E/E' ratio (change from baseline (V1) to 12-week follow-up (V4))
Difference in left ventricular ejection fraction (LVEF) from baseline to 12-week follow-up (V4) | 12 weeks
  Difference in LVEF (systolic function) from baseline to 12-week follow-up
Difference in quality of life (change from baseline to 12-week follow-up) | 12 weeks
  Difference in quality of life from baseline to 12-week follow-up (measured with The Kansas City Cardiomyopathy Questionnaire (KCCQ))
Difference in heart rate variability (HRV) (change from baseline to 12-week follow-up) | 12 weeks
  Difference in HRV from baseline to 12-week follow-up (measured with 24-hour Holter ECG)
Difference in peak VO2 (change from baseline to 12-week follow-up) | 12 weeks
  Difference in peak VO2 from baseline to 12-week follow-up (cardiopulmonary exercise testing)
Change in daily non-sedentary daytime activity from baseline to 12-week follow-up | 12 weeks
  Change in daily non-sedentary daytime activity from baseline to 12-week follow-up (composite measure of movement and locomotion as measured by the Dynaport MoveMonitor) (V4)
Difference in gait speed (change from baseline to 12-week follow-up) | 12 weeks
  Change in gait speed from baseline to 12-week follow-up
Difference in NT-proBNP from baseline to 12-week follow-up | 12 weeks
  Difference in the serum concentration of N-terminal brain natriuretic peptide (NT-proBNP) from baseline to 12-week follow-up
Difference in FEV1 (change from baseline to 12-week follow-up) | 12 weeks
  Difference in forced expiratory volume in one second (FEV1) from baseline to 12-week follow-up
Difference in the augmentation index (change from baseline to 12-week follow-up) | 12 weeks
  Difference in the augmentation index from baseline to 12-week follow-up. The augmentation index is an indicator of arterial stiffness; higher values indicate a worse outcome
Correlations of gait speed | 12 weeks
  Correlations of gait speed during an intermittent supervised test to data assessed in patients' home environment
Difference in METs (change from baseline to 12-week follow-up) | 12 weeks
  Change in metabolic equivalents (METs) from baseline to 12-week follow-up
Difference in daily step count between the intervention groups (change from baseline to 12-week follow-up) | 12 weeks
  Difference in daily step count from baseline to end of study (comparing the two intervention groups only)

OTHER OUTCOMES:
Difference in biomarkers of autonomic function (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of autonomic function from baseline to 6-week follow-up (e.g. heart rate variability)
Difference in biomarkers of autonomic function (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of autonomic function from baseline to 12-week follow-up (e.g. heart rate variability)
Difference in biomarkers of heart failure (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of heart failure from baseline to 6-week follow-up (e.g., NT-proBNP)
Difference in biomarkers of heart failure (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of heart failure from baseline to 12-week follow-up (e.g., NT-proBNP)
Difference in biomarkers of cardio-vascular diseases (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of cardiovascular diseases from baseline to 6-week follow-up (e.g., troponin)
Difference in biomarkers of cardio-vascular diseases (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of cardiovascular diseases from baseline to 12-week follow-up (e.g., troponin)
Difference in biomarkers of metabolic diseases (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of metabolic diseases from baseline to 6-week follow-up (e.g., HbA1c)
Difference in biomarkers of metabolic diseases (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of metabolic diseases from baseline to 12-week follow-up (e.g., HbA1c)
Difference in biomarkers of renal diseases (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of renal diseases from baseline to 6-week follow-up (e.g., eGFR)
Difference in biomarkers of renal diseases (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of renal diseases from baseline to 12-week follow-up (e.g., eGFR)
Difference in biomarkers of cancer (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of cancer from baseline to 6-week follow-up (e.g., LDH)
Difference in biomarkers of cancer (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of cancer from baseline to 12-week follow-up (e.g., LDH)
Difference in biomarkers of pulmonary diseases (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of pulmonary diseases from baseline to 6-week follow-up (e.g., FEV1)
Difference in biomarkers of pulmonary diseases (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of pulmonary diseases from baseline to 12-week follow-up (e.g., FEV1)
Difference in biomarkers of inflammation (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of inflammation from baseline to 6-week follow-up (e.g., C-reactive protein)
Difference in biomarkers of inflammation (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of inflammation from baseline to 12-week follow-up (e.g., C-reactive protein)
Difference in biomarkers of immunity (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of immunity from baseline to 6-week follow-up (e.g., leukocytes)
Difference in biomarkers of immunity (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of immunity from baseline to 12-week follow-up (e.g., leukocytes)
Difference in biomarkers of oxidative stress (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of oxidative stress from baseline to 6-week follow-up (e.g., monocytes)
Difference in biomarkers of oxidative stress (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of oxidative stress from baseline to 12-week follow-up (e.g., monoytes)
Difference in biomarkers of hypercoagulability (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of hypercoagulability from baseline to 6-week follow-up (e.g. mean platelet volume)
Difference in biomarkers of hypercoagulability (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of hypercoagulability from baseline to 12-week follow-up (e.g., mean platelet volume)
Difference in biomarkers of vascular/endothelial function (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of vascular/endothelial function from baseline to 6-week follow-up (e.g. pulse-wave velocity)
Difference in biomarkers of vascular/endothelial function (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of vascular/endothelial function from baseline to 12-week follow-up (e.g. pulse-wave velocity)
Difference in biomarkers of carotid atherosclerosis (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of carotid atherosclerosis from baseline to 6-week follow-up (e.g., intima-media-thickness)
Difference in biomarkers of carotid atherosclerosis (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of carotid atherosclerosis from baseline to 12-week follow-up (e.g., intima-media-thickness)
Difference in biomarkers of methylation (change from baseline to 6-week follow-up) | 6 weeks
  Difference in biomarkers of methylation from baseline to 6-week follow-up (e.g., CpG methylation)
Difference in biomarkers of methylation (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of methylation from baseline to 12-week follow-up (e.g., CpG methylation)
Difference in anthropometrics (change from baseline to 6-week follow-up) | 6 weeks
  Difference in anthropometrics from baseline to 6-week follow-up (e.g., BMI)
Difference in anthropometrics (change from baseline to 12-week follow-up) | 12 weeks
  Difference in anthropometrics from baseline to 12-week follow-up (e.g., BMI)
Difference in biomarkers of psychosomatic diseases (change from baseline to 12-week follow-up) | 12 weeks
  Difference in biomarkers of psychosomatic diseases from baseline to 12-week follow-up (e.g, PHQ-9)
Difference in biomarkers of physical activity | 12 weeks
  Difference in biomarkers of physical activity (e.g., step count)
Difference in biomarkers of sedentary daytime activities | 12 weeks
  Difference in biomarkers of sedentary daytime activities (e.g., sleeping time)
Differences in accelerometry | 12 weeks
  Differences in accelerometry (e.g., measured with the Dynaport MoveMonitor)
Evaluation of compliance of study participants with the mobile devices | 12 weeks
  Explorative evaluation of compliance as assessed with technical data from the mobile devices (e.g. wearing time) and a qualitative questionnaire on device experience (allowing to evaluate inter alia feasibility and wearability)
Evaluation of functionality of the mobile devices | 12 weeks
  Explorative evaluation of device functionality (e.g., as measured by number of data points per observation period)
Evaluation of realibility of the mobile devices | 12 weeks
  Explorative evaluation of realibility of mobile device measurements (e.g. by comparing systolic blood pressure measurements between mobile devices and routine measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Wild, Univ.-Prof. Dr. med., MSc, Principal Investigator — University Medical Center Mainz
Locations (1):
- University Medical Center of the Johannes Gutenberg-University Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeid S, Prochaska JH, Schuch A, Trobs SO, Schulz A, Munzel T, Pies T, Dinh W, Michal M, Simon P, Wild PS. Personalized app-based coaching for improving physical activity in heart failure with preserved ejection fraction patients compared with standard care: rationale and design of the MyoMobile Study. Eur Heart J Digit Health. 2025 Jan 30;6(2):298-309. doi: 10.1093/ehjdh/ztae096. eCollection 2025 Mar. PMID 40110212